CLINICAL TRIAL: NCT02547012
Title: Comparison of Two Rescue Therapies for Helicobacter Pylori Infection - A Multicenter Randomized Controlled Trial
Brief Title: Comparison of Two Rescue Therapies for Helicobacter Pylori Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS13-CT11-15
Record Dates: First submitted 2015-09-06; First posted 2015-09-11 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Eradication rate; Rescue treatment
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Levofloxacin; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- esomeprazole+amox+levo+tetra (Experimental): esomeprazole 40 mg b.d., amoxicillin 500 mg q.d.s., levofloxacin 500 mg o.d., and tetracycline 500 mg q.d.s.
  Interventions: Drug: esomeprazole+amox+levo+tetra
- esomeprazole+amox+levo (Active Comparator): esomeprazole 40 mg b.d., amoxicillin 500 mg q.d.s., and levofloxacin 500 mg o.d.
  Interventions: Drug: esomeprazole+amox+levo

INTERVENTIONS:
Drug: esomeprazole+amox+levo+tetra — esomeprazole 40 mg b.d., amoxicillin 500 mg q.d.s., levofloxacin 500 mg o.d., and tetracycline 500 mg q.d.s.
  Other Names: esomeprazole 40mg; amoxicillin 500 mg; levofloxacin 500 mg; tetracycline 500 mg
  Arms: esomeprazole+amox+levo+tetra
Drug: esomeprazole+amox+levo — esomeprazole 40 mg b.d., amoxicillin 500 mg q.d.s., levofloxacin 500 mg o.d.,
  Other Names: esomeprazole 40 mg; amoxicillin 500 mg; levofloxacin 500 mg
  Arms: esomeprazole+amox+levo

SUMMARY:
From the profiles of antibiotic susceptibility data following eradication therapy, tetracycline, amoxicillin and levofloxacin are all good candidates of antibiotics used in the rescue treatment.

DETAILED DESCRIPTION:
The H pylori-infected adult patients with failure of standard triple therapy and H pylori-infected adult patients with failure of non-bismuth quadruple therapy are randomly assigned to either EALT (esomeprazole 40 mg b.d., amoxicillin 500 mg q.d.s., levofloxacin 500 mg o.d., and tetracycline 500 mg q.d.s.) therapy or EAL (esomeprazole 40 mg b.d., amoxicillin 500 mg q.d.s., and levofloxacin 500 mg o.d.) for 10 days. Repeated endoscopy with rapid urease test, histological examination and culture or urea breath tests is performed at six weeks after the end of anti-H pylori therapy.

ELIGIBILITY:
Inclusion Criteria:

* positive results of both rapid urease test and histology,
* a positive result of urea breath test,
* or a positive result of culture.

Exclusion Criteria:

* ingestion of antibiotics, bismuth, or proton pump inhibitor（PPI）within the prior 4 weeks,
* patients with allergic history to the medications used,
* patients with previous gastric surgery,
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia),
* pregnant women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-11; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Suerbaum S, Michetti P. Helicobacter pylori infection. N Engl J Med. 2002 Oct 10;347(15):1175-86. doi: 10.1056/NEJMra020542. No abstract available. PMID 12374879
- [Background] Malfertheiner P, Chan FK, McColl KE. Peptic ulcer disease. Lancet. 2009 Oct 24;374(9699):1449-61. doi: 10.1016/S0140-6736(09)60938-7. Epub 2009 Aug 13. PMID 19683340
- [Background] Sung JJ, Chung SC, Ling TK, Yung MY, Leung VK, Ng EK, Li MK, Cheng AF, Li AK. Antibacterial treatment of gastric ulcers associated with Helicobacter pylori. N Engl J Med. 1995 Jan 19;332(3):139-42. doi: 10.1056/NEJM199501193320302. PMID 7800005
- [Background] Zucca E, Dreyling M; ESMO Guidelines Working Group. Gastric marginal zone lymphoma of MALT type: ESMO clinical recommendations for diagnosis, treatment and follow-up. Ann Oncol. 2009 May;20 Suppl 4:113-4. doi: 10.1093/annonc/mdp146. No abstract available. PMID 19454427
- [Background] Asaka M, Kato M, Takahashi S, Fukuda Y, Sugiyama T, Ota H, Uemura N, Murakami K, Satoh K, Sugano K; Japanese Society for Helicobacter Research. Guidelines for the management of Helicobacter pylori infection in Japan: 2009 revised edition. Helicobacter. 2010 Feb;15(1):1-20. doi: 10.1111/j.1523-5378.2009.00738.x. PMID 20302585
- [Background] Malfertheiner P, Megraud F, O'Morain C, Bazzoli F, El-Omar E, Graham D, Hunt R, Rokkas T, Vakil N, Kuipers EJ. Current concepts in the management of Helicobacter pylori infection: the Maastricht III Consensus Report. Gut. 2007 Jun;56(6):772-81. doi: 10.1136/gut.2006.101634. Epub 2006 Dec 14. PMID 17170018
- [Background] Fock KM, Katelaris P, Sugano K, Ang TL, Hunt R, Talley NJ, Lam SK, Xiao SD, Tan HJ, Wu CY, Jung HC, Hoang BH, Kachintorn U, Goh KL, Chiba T, Rani AA; Second Asia-Pacific Conference. Second Asia-Pacific Consensus Guidelines for Helicobacter pylori infection. J Gastroenterol Hepatol. 2009 Oct;24(10):1587-600. doi: 10.1111/j.1440-1746.2009.05982.x. PMID 19788600
- [Background] Graham DY, Fischbach L. Helicobacter pylori treatment in the era of increasing antibiotic resistance. Gut. 2010 Aug;59(8):1143-53. doi: 10.1136/gut.2009.192757. Epub 2010 Jun 4. PMID 20525969
- [Background] Gumurdulu Y, Serin E, Ozer B, Kayaselcuk F, Ozsahin K, Cosar AM, Gursoy M, Gur G, Yilmaz U, Boyacioglu S. Low eradication rate of Helicobacter pylori with triple 7-14 days and quadriple therapy in Turkey. World J Gastroenterol. 2004 Mar 1;10(5):668-71. doi: 10.3748/wjg.v10.i5.668. PMID 14991935
- [Background] Bigard MA, Delchier JC, Riachi G, Thibault P, Barthelemy P. One-week triple therapy using omeprazole, amoxycillin and clarithromycin for the eradication of Helicobacter pylori in patients with non-ulcer dyspepsia: influence of dosage of omeprazole and clarithromycin. Aliment Pharmacol Ther. 1998 Apr;12(4):383-8. doi: 10.1046/j.1365-2036.1998.00315.x. PMID 9690730
- [Background] Gatta L, Vakil N, Leandro G, Di Mario F, Vaira D. Sequential therapy or triple therapy for Helicobacter pylori infection: systematic review and meta-analysis of randomized controlled trials in adults and children. Am J Gastroenterol. 2009 Dec;104(12):3069-79; quiz 1080. doi: 10.1038/ajg.2009.555. Epub 2009 Oct 20. PMID 19844205
- [Background] Chuah SK, Tsay FW, Hsu PI, Wu DC. A new look at anti-Helicobacter pylori therapy. World J Gastroenterol. 2011 Sep 21;17(35):3971-5. doi: 10.3748/wjg.v17.i35.3971. PMID 22046084
- [Background] Wu DC, Hsu PI, Wu JY, Opekun AR, Kuo CH, Wu IC, Wang SS, Chen A, Hung WC, Graham DY. Sequential and concomitant therapy with four drugs is equally effective for eradication of H pylori infection. Clin Gastroenterol Hepatol. 2010 Jan;8(1):36-41.e1. doi: 10.1016/j.cgh.2009.09.030. Epub 2009 Oct 3. PMID 19804842
- [Background] Hsu PI, Wu DC, Wu JY, Graham DY. Modified sequential Helicobacter pylori therapy: proton pump inhibitor and amoxicillin for 14 days with clarithromycin and metronidazole added as a quadruple (hybrid) therapy for the final 7 days. Helicobacter. 2011 Apr;16(2):139-45. doi: 10.1111/j.1523-5378.2011.00828.x. PMID 21435092
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Wu DC, Hsu PI, Tseng HH, Tsay FW, Lai KH, Kuo CH, Wang SW, Chen A. Helicobacter pylori infection: a randomized, controlled study comparing 2 rescue therapies after failure of standard triple therapies. Medicine (Baltimore). 2011 May;90(3):180-185. doi: 10.1097/MD.0b013e31821c9d1c. PMID 21512411
- [Background] Gisbert JP. "Rescue" regimens after Helicobacter pylori treatment failure. World J Gastroenterol. 2008 Sep 21;14(35):5385-402. doi: 10.3748/wjg.14.5385. PMID 18803350
- [Background] Hojo M, Miwa H, Nagahara A, Sato N. Pooled analysis on the efficacy of the second-line treatment regimens for Helicobacter pylori infection. Scand J Gastroenterol. 2001 Jul;36(7):690-700. doi: 10.1080/003655201300191941. PMID 11444467
- [Background] Saad RJ, Schoenfeld P, Kim HM, Chey WD. Levofloxacin-based triple therapy versus bismuth-based quadruple therapy for persistent Helicobacter pylori infection: a meta-analysis. Am J Gastroenterol. 2006 Mar;101(3):488-96. doi: 10.1111/j.1572-0241.2006.00637.x. PMID 16542284
- [Background] Kuo CH, Hu HM, Kuo FC, Hsu PI, Chen A, Yu FJ, Tsai PY, Wu IC, Wang SW, Li CJ, Weng BC, Chang LL, Jan CM, Wang WM, Wu DC. Efficacy of levofloxacin-based rescue therapy for Helicobacter pylori infection after standard triple therapy: a randomized controlled trial. J Antimicrob Chemother. 2009 May;63(5):1017-24. doi: 10.1093/jac/dkp034. Epub 2009 Feb 26. PMID 19246508
- [Background] Pontone S, Standoli M, Angelini R, Pontone P. Efficacy of H. pylori eradication with a sequential regimen followed by rescue therapy in clinical practice. Dig Liver Dis. 2010 Aug;42(8):541-3. doi: 10.1016/j.dld.2009.12.007. Epub 2010 Jan 12. PMID 20061196
- [Background] Manfredi M, Bizzarri B, de'Angelis GL. Helicobacter pylori infection: sequential therapy followed by levofloxacin-containing triple therapy provides a good cumulative eradication rate. Helicobacter. 2012 Aug;17(4):246-53. doi: 10.1111/j.1523-5378.2012.00945.x. Epub 2012 Mar 20. PMID 22759323
- [Background] Perna F, Zullo A, Ricci C, Hassan C, Morini S, Vaira D. Levofloxacin-based triple therapy for Helicobacter pylori re-treatment: role of bacterial resistance. Dig Liver Dis. 2007 Nov;39(11):1001-5. doi: 10.1016/j.dld.2007.06.016. Epub 2007 Sep 21. PMID 17889627
- [Background] Zullo A, Scaccianoce G, De Francesco V, Ruggiero V, D'Ambrosio P, Castorani L, Bonfrate L, Vannella L, Hassan C, Portincasa P. Concomitant, sequential, and hybrid therapy for H. pylori eradication: a pilot study. Clin Res Hepatol Gastroenterol. 2013 Dec;37(6):647-50. doi: 10.1016/j.clinre.2013.04.003. Epub 2013 Jun 6. PMID 23747131
- [Background] Gisbert JP, Molina-Infante J, Marin AC, Vinagre G, Barrio J, McNicholl AG. Second-line rescue triple therapy with levofloxacin after failure of non-bismuth quadruple "sequential" or "concomitant" treatment to eradicate H. pylori infection. Scand J Gastroenterol. 2013 Jun;48(6):652-6. doi: 10.3109/00365521.2013.786132. Epub 2013 Apr 5. PMID 23556551
- [Background] Hsu PI, Lai KH, Tseng HH, Lo GH, Lo CC, Lin CK, Cheng JS, Chan HH, Ku MK, Peng NJ, Chien EJ, Chen W, Hsu PN. Eradication of Helicobacter pylori prevents ulcer development in patients with ulcer-like functional dyspepsia. Aliment Pharmacol Ther. 2001 Feb;15(2):195-201. doi: 10.1046/j.1365-2036.2001.00903.x. PMID 11148437
- [Background] Hsu PI, Lai KH, Tseng HH, Liu YC, Yen MY, Lin CK, Lo GH, Huang RL, Huang JS, Cheng JS, Huang WK, Ger LP, Chen W, Hsu PN. Correlation of serum immunoglobulin G Helicobacter pylori antibody titers with histologic and endoscopic findings in patients with dyspepsia. J Clin Gastroenterol. 1997 Dec;25(4):587-91. doi: 10.1097/00004836-199712000-00007. PMID 9451668
- [Background] Hsu PI, Lai KH, Chien EJ, Lin CK, Lo GH, Jou HS, Cheng JS, Chan HH, Hsu JH, Ger LP, Hsu PN, Tseng HH. Impact of bacterial eradication on the cell proliferation and p53 protein accumulation in Helicobacter pylori-associated gastritis. Anticancer Res. 2000 Mar-Apr;20(2B):1221-8. PMID 10810425
- [Background] Peng NJ, Lai KH, Liu RS, Lee SC, Tsay DG, Lo CC, Tseng HH, Huang WK, Lo GH, Hsu PI. Endoscopic 13C-urea breath test for the diagnosis of Helicobacter pylori infection. Dig Liver Dis. 2003 Feb;35(2):73-7. doi: 10.1016/s1590-8658(03)00014-8. PMID 12747623
- [Background] Peng NJ, Lai KH, Liu RS, Lee SC, Tsay DG, Lo CC, Tseng HH, Huang WK, Lo GH, Hsu PI. Clinical significance of oral urease in diagnosis of Helicobacter pylori infection by [13C]urea breath test. Dig Dis Sci. 2001 Aug;46(8):1772-8. doi: 10.1023/a:1010626225949. PMID 11508681
- [Background] Kita T, Sakaeda T, Aoyama N, Sakai T, Kawahara Y, Kasuga M, Okumura K. Optimal dose of omeprazole for CYP2C19 extensive metabolizers in anti-Helicobacter pylori therapy: pharmacokinetic considerations. Biol Pharm Bull. 2002 Jul;25(7):923-7. doi: 10.1248/bpb.25.923. PMID 12132671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: Oct 2013 - Jul 2017 Type of location: Kaohsiung Veterans General Hospital and Kaohsiung Medical University Chung-Ho Memorial Hospital
Pre-assignment Details: None were excluded following participant enrollment.
Period: Overall Study
Arm/Group | Esomeprazole+Amox+Levo+Tetra | Esomeprazole+Amox+Levo
Started | 24 | 27
Completed | 24 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole+Amox+Levo+Tetra | Esomeprazole+Amox+Levo | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.88 (9.13) | 56.44 (15.02) | 56.79 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 27 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 24 | 27 | 51
history of smoking [Number; unit: participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Which H. Pylori Was Eradicated
Description: Evaluate eradication outcome by endoscopy urease test and histology or urea breath test
Time Frame: six weeks after the end of anti-H pylori therapy.
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Esomeprazole+Amox+Levo+Tetra | Esomeprazole+Amox+Levo
Number analyzed (Participants) | 24 | 27
participants | 13 | 21

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Esomeprazole+Amox+Levo+Tetra | Esomeprazole+Amox+Levo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 14/24 | 5/27
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esomeprazole+Amox+Levo+Tetra (N=24) | Esomeprazole+Amox+Levo (N=27)
Nausea (Gastrointestinal disorders) | 12 (12) | 2 (2) — Patients had Nausea discomforts.
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) — Patients had dizziness discomforts.

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT02547012/Prot_SAP_000.pdf